CLINICAL TRIAL: NCT06761326
Title: Right Versus Left Ultrasound-Guided Distal Axillary Approach For Subclavian Vein Cannulation : A Prospective Randomized Pilot Study
Brief Title: Right Versus Left Distal Axillary Approach For Subclavian Vein Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Engi Yousry, Lecturer of anesthesia and pain medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Axillary subclavian approach
Record Dates: First submitted 2024-10-10; First posted 2025-01-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-01

CONDITIONS: Infraclavicular Vein Cannulation; Venous Cannulation
Keywords: subclavian vein cannulation; ultrasound guided; fluroscopy; maldirection; infraclavicular approach

STUDY DESIGN:
Intervention Model Description: A randomized controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right subclavian vein cannulation (Other): All patients will be in supine position, with the right arm abducted to 45 degrees , the angle of the arm will be increased to 90 degrees to best acquire the image. The probe will be placed in he parasagittal plane in the deltopectoral groove of the right side , medial to the coracoid process . The image will be optimized for the best image of the right axillary artery and vein similar to that acquired when performing an infraclavicular approach for brachial plexus block . The probe will be rotated to obtain a longitudinal image of the right axillary vein . The needle will be introduced in real time imaging , in an in plane technique and blood will be aspirated , the guidewire will be introduced in real time imaging. The internal jugular vein will be scanned bilaterally via ultrasonography to exclude malposition of the guidewire and will be reported in case of such. The catheter will be introduced through the sheath and will be tunneled the skin.
  Interventions: Procedure: Ultrasound guided right infraclavicular approach of subclavian vein cannulation
- Left subclavian vein cannulation (Experimental): All patients will be in supine position, with the left arm abducted to 45 degrees , the angle of the arm will be increased to 90 degrees to best acquire the image. The probe will be placed in he parasagittal plane in the left deltopectoral groove medial to the coracoid process . The image will be optimized regarding the depth , focus and the gain accordingly for the best image of the axillary artery and vein similar to that acquired when performing an infraclavicular approach for brachial plexus block . The probe will be rotated to obtain a longitudinal image of the left axillary vein . The needle will be introduced in real time imaging , in an in plane technique and blood will be aspirated , the guidewire will be introduced in real time imaging. The internal jugular vein will be scanned bilaterally via ultrasonography to exclude malposition of the guidewire and will be reported in case of such. The catheter will be introduced through the sheath and will be tunneled the skin.
  Interventions: Procedure: Ultrasound guided left infraclavicular approach of subclavian vein cannulation

INTERVENTIONS:
Procedure: Ultrasound guided right infraclavicular approach of subclavian vein cannulation — All patients will be in supine position, with the arm abducted to 45 degrees , the angle of the arm will be increased to 90 degrees to best acquire the image.The probe will be placed in he parasgittal plane in the deltopectoral groove medial to the coracoid process . The image will be optimized regarding the depth , focus and the gain accorgingly for the best image of the axillary artery and vein similar to that acquired when performing an infraclavicular approach for brachial plexus block . The probe will be rotated to obtain a longitudinal image of the axillary vein . The needle will be introduced in real time imaging , in an inplane technique and blood will be aspirated , the guidewire will be introduced in real time imaging.The internal jugular vein will be scanned bilaterally via ultrasonography to exclude malposition of the guidewire and will be reported in case of such. The catheter will be introduced through the sheath and will be tunneled the skin.
  Arms: Right subclavian vein cannulation
Procedure: Ultrasound guided left infraclavicular approach of subclavian vein cannulation — All patients will be in supine position, with the arm abducted to 45 degrees , the angle of the arm will be increased to 90 degrees to best acquire the image.The probe will be placed in he parasgittal plane in the deltopectoral groove medial to the coracoid process . The image will be optimized regarding the depth , focus and the gain accorgingly for the best image of the axillary artery and vein similar to that acquired when performing an infraclavicular approach for brachial plexus block . The probe will be rotated to obtain a longitudinal image of the axillary vein . The needle will be introduced in real time imaging , in an inplane technique and blood will be aspirated , the guidewire will be introduced in real time imaging.The internal jugular vein will be scanned bilaterally via ultrasonography to exclude malposition of the guidewire and will be reported in case of such. The catheter will be introduced through the sheath and will be tunneled the skin.
  Arms: Left subclavian vein cannulation

SUMMARY:
Central venous cannulation is an essential procedure in the anaesthetic and critical care practice. Ultrasound has revolutionized the practice favoring the internal jugular cannulation to the other sites .Subcalvian vein cannulation has fallen out of favor mainly due to the difficult visualization with the ultrasound, especially in obese patients and the inevitable position of the clavicle acting as a bony obstacle , in addition to the anatomical position in vicinity to the pleura which might raise the risk of pneumothorax . Indeed the subclavian vein cannulation is more comfortable and tolerated by the patient especially those requiring long term intravenous therapy, with less rates of infection and thrombosis. This mandated the development of a safer and efficient technique for the cannulation empowered by the ultrasound technology.

The infracalvicular approach or the proximal axillary vein cannulation has been described but is not popular. It provides a potentially safer and successful technique with less complication both in "experienced" and "less experienced"operators . All the patients will receive general anaesthesia with laryngeal mask insertion . Careful sterilization of the surgical site and strict aseptic techniques for the handling of the ultrasound probe will be pursued

DETAILED DESCRIPTION:
All patients will be in supine position, with the arm abducted to 45 degrees , the angle of the arm will be adjusted to acquire best image. The probe will be placed in he parasagittal plane in the deltopectoral groove medial to the coracoid process . The image will be optimized regarding the depth , focus and the gain accordingly for the best image of the axillary artery and vein similar to that acquired when performing an infraclavicular approach for brachial plexus block . The probe will be rotated to obtain a longitudinal image of the axillary vein . The needle will be introduced in real time imaging , in an in-plane technique and blood will be aspirated , the guidewire will be introduced in real time imaging .The internal jugular vein will be scanned bilaterally via ultrasonography to exclude malposition of the guidewire and will be reported in case of such. The catheter will be introduced through the sheath and will be tunneled the skin, Infraclavicular incision will be performed for the port site , the port will be secured in a dissected pocket right above the pectoralis major muscle .Flush back will be confirmed from the port .The incision will be closed in layers .The final position of the catheter tip will be confirmed using fluoroscopic guidance. In case of difficult visualization or failure of cannulation of one side , the subclavian vein of the contralateral side will be scanned and cannulated . The internal jugular vein will be the cannulated instead if any further difficulties were encountered .

ELIGIBILITY:
Inclusion Criteria:

.Patients requiring porta Cath insertion.

Exclusion Criteria:

* Abnormalities in the platelet count or coagulation
* Thrombosis of the target vein
* Soft tissue infection of the overlying area
* Fracture of the clavicle or proximal ribs
* Patients with pacemakers or defibrillators
* Malignant superior vena cava syndrome
* Gross obesity
* History of prior catheterization of the subclavian vein
* Patient refusal to participate in the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Successful cannulation | Directly after the end of the procedure
  Recognition of the catheter in the SVC by fluoroscopy

SECONDARY OUTCOMES:
Rate of malposition identified by the ultrasound | Directly after the insertion of the guidewire and the catheter
  The ultrasound probe will be positioned on the internal jugular vein for the recognition of malposition of the guidewire
Complication of the procedures | Directly at the end of the procedure
  All the complications will be recognized and reported

CONTACTS AND LOCATIONS:
Overall Officials: Engi Y Hashem, MD, Principal Investigator — Medical research institute , Alexandria university
Locations (1):
- Medical Research Institute, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
unfortunately there is no web site for the publication of results , but whoever is interested in the study can contact the main author

REFERENCES:
- [Background] Kim YJ, Ma S, Yoon HK, Lee HC, Park HP, Oh H. Supraclavicular versus infraclavicular approach for ultrasound-guided right subclavian venous catheterisation: a randomised controlled non-inferiority trial. Anaesthesia. 2022 Jan;77(1):59-65. doi: 10.1111/anae.15525. Epub 2021 Jul 6. PMID 34231204
- [Background] Imai E, Watanabe J, Okano H, Yokozuka M. Efficacy and safety of supraclavicular versus infraclavicular approach for subclavian vein catheterisation: An updated systematic review and meta-analysis of randomised controlled trials. Indian J Anaesth. 2023 Jun;67(6):486-496. doi: 10.4103/ija.ija_837_22. Epub 2023 Jun 14. PMID 37476443
- [Background] Hosur Ravikumar R, Majage S, Prasanna M, Ray BR. Comparison of ultrasound guided supraclavicular subclavian vein versus infraclavicular subclavian/axillary vein catheterization: A systematic review and meta analysis. J Vasc Access. 2025 Mar;26(2):633-640. doi: 10.1177/11297298241239092. Epub 2024 Mar 20. PMID 38506879